CLINICAL TRIAL: NCT01524744
Title: A Randomized Clinical Trial of the Effect of Pimecrolimus Cream 1% Compared With Topical Corticosteroid in Treatment of Erosive Oral Lichen Planus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, ATESSA PAKFETRAT, Associate professor, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 87909; 87909 (Other: 87909)
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Oral Lichen Planus
Keywords: oral lichen planus treatment pimecrolimus
MeSH Terms: conditions — Lichen Planus, Oral | interventions — Gramicidin, Neomycin Sulfate, Nystatin, Triamcinolone Acetonide Drug Combination

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pimecrolimus ointment 0.1 % (Active Comparator): This group used drugs 3 times a day for 2 months and then didn't eat or drink for 20 minutes after use
  Interventions: Drug: Pimecrolimus ointment; Drug: Adcortyl
- Adcortyle (Active Comparator): Control group used adcortyle (triamcinolone acetonide 0.1% in orabase, Bristol-Myers Squibbb, Anagn, Italy)
  Interventions: Drug: Adcortyl

INTERVENTIONS:
Drug: Pimecrolimus ointment — Case group used drugs 3 times a day for 2 months and then didn't eat or drink for 20 minutes after use
  Arms: Pimecrolimus ointment 0.1 %
Drug: Adcortyl — triamcinolone acetonide 0.1% in orabase

SUMMARY:
The purpose of this study is to compare the effect of topical Pimecrolimus with adcortyl on erosive-atrophic 0ral lichen planus in a randomized clinical trial study.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed oral lichen planus in combination with a compatible clinical appearance was used for diagnosis.

Exclusion Criteria:

* Unable to undergo oral biopsy for diagnosis
* Systemic diseases or malignancy
* Pregnancy
* Lesion/lesions with dysplasia/ history of allergic reaction to corticosteroids or immunomodulatory drugs.
* Lesions adjacent to amalgam filling were also excluded from this study.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-03; Primary Completion 2012-10 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
signs of oral lichen planus | every 2 weeks
  size and type of oral lichen planus has been recorded

SECONDARY OUTCOMES:
symptoms of oral lichen planus | every 2 weeks
  pain of oral lesions has been recorded

CONTACTS AND LOCATIONS:
Overall Officials: atessa pakfetrat, associate professor, Principal Investigator — Mashhad University of Medical Science
Locations (1):
- Mashhad University of Medical Science, Mashhad, Khorasan Razavi, Iran